CLINICAL TRIAL: NCT05313568
Title: Instant Effect of Self Stretching, Plantar Self Massage and Manual Stimulation on Balance and Reaction Time in Healthy Individuals
Brief Title: Self Stretching, Plantar Self Massage and Manual Stimulation on Balance and Reaction Time
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Miray Budak, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Foot.Balance.ReactionTime.
Record Dates: First submitted 2021-10-14; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Healthy; Stretch
Keywords: Self Stretching, Self Massage, Manual Stimulation, Balance, Reaction Time, Healthy
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- static stretching group (Active Comparator): The stretch will be done by placing both feet on a raised platform, lowering the heel off the platform without touching the ground, and held in this position to perform a static stretch. They will perform 5 repetitions, 15 seconds of rest and 1 minute of stretching.
  Interventions: Other: static stretching
- self massage group (Experimental): In addition to the self-stretching application, plantar self-massage will be applied. Plantar self massage will be shown to the participants by the physiotherapist with a 7 cm spiky massage ball. Then, participants will be asked to self-massage the plantar sole of the foot for 5 minutes with a 7 cm spiky massage ball.
  Interventions: Other: static stretching; Other: self massage
- Manual Stimulation Group (Experimental): In addition to the self-stretching application, manual stimulation will be applied.
  Manual protocol:
  A) Pressure will be applied in each interdigital space and on the longitudinal arch with shear in the longitudinal direction (5 repetitions of 10 seconds each).
  B) Pressure with transverse shear on the metatarsal heads (5 repetitions of 5 seconds each) C) Static pressure will be applied to the first and fifth metatarsal head, center of the midfoot, and heel (5 repetitions per 10-second period each).
  Interventions: Other: static stretching; Other: Manual Stimulation

INTERVENTIONS:
Other: static stretching — The stretch will be done by placing both feet on a raised platform, lowering the heel off the platform without touching the ground, and held in this position to perform a static stretch. They will perform 5 repetitions, 15 seconds of rest and 1 minute of stretching.
Other: self massage — In addition to the self-stretching application, plantar self-massage will be applied. Plantar self massage will be shown to the participants by the physiotherapist with a 7 cm spiky massage ball. Then, participants will be asked to self-massage the plantar sole of the foot for 5 minutes with a 7 cm spiky massage ball.
  Arms: self massage group
Other: Manual Stimulation — In addition to the self-stretching application, manual stimulation will be applied.
  Manual protocol:
  A) Pressure will be applied in each interdigital space and on the longitudinal arch with shear in the longitudinal direction (5 repetitions of 10 seconds each).
  B) Pressure with transverse shear on the metatarsal heads (5 repetitions of 5 seconds each) C) Static pressure will be applied to the first and fifth metatarsal head, center of the midfoot, and heel (5 repetitions per 10-second period each).
  Arms: Manual Stimulation Group

SUMMARY:
The aim of this study is to investigate the instantaneous effects of self-stretching, plantar self-massage and manual stimulation on balance and reaction time in healthy individuals. 102 individuals meeting the inclusion criteria will be included in the study. Individuals will be randomly divided into 3 groups: static stretching group (n=34), self-massage group (n=34) and manual stimulation group (n=34). Static stretching will be applied to all individuals (n=102). In addition to static stretching, self-massage will be applied to individuals in the self-massage group (n=34). Individuals in the manual stimulation group (n=34) will receive manual stimulation in addition to static stretching. Individuals will be evaluated in terms of static balance, dynamic balance, reaction time and foot functionality before and immediately after the applications.

ELIGIBILITY:
Inclusion Criteria:

* being between 18 and 50 years old
* having Body Mass Index (BMI) limit to be 20-25
* having Normal range of motion of the ankle joint
* having the score of the foot is between 0 and +5 according to the foot posture index,
* having the score 3+ on ankle muscle strength

Exclusion Criteria:

* being pregnant
* having undergone surgery on the foot and ankle in the last 6 months
* history of lower extremity injury with residual symptoms in the past year
* having diseases that affect the balance such as rheumatic disease, osteoarthritis, multiple sclerosis
* being professional athlete
* presence of vestibular disease (Meniere, Vertigo etc.), diabetes, neuropathy Being in
* being in the menopausal period
* having hip flexor muscle shortening
* having basal ganglia disorders such as Parkinson's disease, Huntington's disease
* having sensory problems on the sole of the foot

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
One Leg Standing Test | change in static balance immediately after application
  It will be used to evaluate static balance. If the cut-off value is <10 seconds, there is a balance disorder, if it is <5 seconds, there is a risk of falling.
Functional Reach Test | change in dynamic balance immediately after application
  It will be used to evaluate dynamic balance. The distance that the person can reach is measured. Higher scores mean better performance.
Y Balance Test | change in dynamic balance immediately after application
  It will be used to evaluate dynamic balance. The distance that the person can reach is measured. Higher scores mean better performance.
Nelson's Foot Reaction Time Test | change in reaction time immediately after application
  It will be used to evaluate reaction time. The time that the person can react is measured. Higher scores mean worse performance.

SECONDARY OUTCOMES:
Active-passive Limb Matching Test | change in proprioception immediately after application
  It will be used to evaluate proprioception. Same position mean better performance.
Goniometer | change in range of motion immediately after application
  It will be used to evaluate range of motion of ankle. Dorsiflexion range of motion is 20 degree. Plantar flexion range of motion is 50 degree. Eversion range of motion is 15 degree. Inversion range of motion is 35 degree. Higher score means better performance.
Foot Posture Index | change in foot posture immediately after application
  It will be used to evaluate foot posture. Palpation of the talus head in the hindfoot, inclination under and over the lateral malleolus, pronation/supination of the calcaneus, ballooning in the talonavicular joint region in the forefoot, medial longitudinal arch structure, and abduction/adduction of the forefoot relative to the hindfoot are evaluated. Each of these criteria takes values between -2 and +2. 0 means the foot is in neutral position, positive values are interpreted as pronation, and negative values are interpreted as supination.
Thomas test | change in hip flexor shortness immediately after application
  It will be used to evaluate hip flexor shortness. If the other leg raise, it is positive.
Pointed-blunt Test | change in sensory immediately after application
  It will be used to evaluate presence of sensory problems. Higher scores mean worse performance.
  Scoring:
  Normal <6mm Fair 6-10mm Poor 11-15mm

CONTACTS AND LOCATIONS:
Overall Officials: Miray BUDAK, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)